CLINICAL TRIAL: NCT06144190
Title: Impact of Discharge Criteria on the Length of Stay in Preterm Infants: a Retrospective Study in Japan and Finland
Brief Title: Discharge Criteria of Preterm Infants
Status: Completed | Type: Observational
Sponsor: Nagano Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryo Itoshima, Chief physician, Nagano Children's Hospital
Other Study IDs: S-04-49
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Length of Stay
Keywords: Early discharge; Family centered care; Tube feeding; Transition to home; Neonatal home care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Japan: Preterm infants born at 28 to 31 gestational weeks in 2020-2021 in a Level IV NICU in Japan
- Finland: Preterm infants born at 28 to 31 gestational weeks in 2020-2021 in a Level III NICU in Finland

SUMMARY:
This retrospective study aims to compare discharge criteria and their impact on the length of stay using two neonatal intensive care units from two countries. The possible discharge criteria include temperature control, apnea observation, periodic respiration, least weight limit, and parents' readiness.

The data were collected retrospectively in each study site.

DETAILED DESCRIPTION:
Aims: To compare discharge criteria and their impact on the length of stay among preterm infants in Japan and Finland. The possible discharge criteria include temperature control, apnea observation, periodic respiration, least weight limit, and parents' readiness.

Study design and settings: This is a retrospective comparison study in two NICUs: a Level IV in Japan and a Level III in Finland.

Patients: Eligible infants are those who were born between 28+0 and 31+6 weeks of gestation and who were discharged home from the study sites between January 2020 and December 2021. Infants will be excluded if (1) they have major anomalies at birth, (2) they are not discharged home from the study sites, or (3) they are discharged home with oxygen and/or after tracheostomy.

Outcome measures: The primary outcomes are the most common last discharge criterion between the two NICUs, and the potential shortening effects of each discharge criterion on the length of stay. The secondary outcome is the postmenstrual age (PMA) for each discharge criterion.

Statistics: The comparison between two continuous variables will be carried out by the student t test.

Ethics: The Ethics Committee of Nagano Children's Hospital gave ethical approval to this study. The study permission was obtained in both study sites.

ELIGIBILITY:
Inclusion Criteria:

* Born between 28 and 31 weeks of gestation and
* Discharged home from the study sites between January 2020 and December 2021

Exclusion Criteria:

* Having major anomalies at birth
* Need for home oxygen therapy, tracheostomy, and/or gastrostomy at discharge

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborns who were born and taken care of in two neonatal intensive care units (NICUs): a Level IV NICU at Nagano Children's Hospital in Japan and a Level III NICU at Turku University Hospital in Finland.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Last discharge criterion | at discharge (about 2 months of age)
  The most common last discharge criterion that was met in each study site
Effects of each discharge criterion on the length of stay | at discharge (about 2 months of age)
  The potential shortening effects of each discharge criterion on the length of stay

SECONDARY OUTCOMES:
The postmenstrual age for each discharge criterion | at discharge (about 2 months of age)
  The postmenstrual age for each discharge criterion that was met

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Itoshima, MD, Principal Investigator — Nagano Children's Hospital; Liisa Lehtonen, MD, Study Director — Turku University Hospital
Locations (1):
- Nagano Children's Hospita, Azumino, Nagano, Japan

IPD SHARING:
Plan to Share IPD: Undecided
It might be possible only after the necessary procedures have been followed including study permissions in both study sites.